CLINICAL TRIAL: NCT02077166
Title: A Multicenter Open-Label Phase 1b/2 Study of the Bruton's Tyrosine Kinase (BTK) Inhibitor, Ibrutinib, in Combination With Lenalidomide and Rituximab in Subjects With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Brief Title: Ibrutinib in Combination With Lenalidomide and Rituximab in Participants With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Collaborators: Janssen Research & Development, LLC (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1123-CA; 2013-004341-17 (EudraCT Number)
Record Dates: First submitted 2014-02-10; First posted 2014-03-04 (Estimated); Results first posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Relapsed Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma
Keywords: DLBCL
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — ibrutinib; Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Phase 1b: Enrolled at Lenalidomide Dose 15 mg (Dose Level 1) (Experimental): Ibrutinib 560 mg administered orally (PO) once daily (QD) beginning Cycle 1 Day 1 until disease progression or unacceptable toxicity. Lenalidomide 15 mg administered PO QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity. Rituximab 375 mg/m^2 administered intravenously (IV) on Day 1 of each 28-day cycle for 6 cycles.
  Interventions: Drug: Ibrutinib; Drug: Lenalidomide; Drug: Rituximab
- Phase 1b: Enrolled at Lenalidomide Dose 10 mg (Dose Level -1) (Experimental): De-escalation cohort: Ibrutinib 560 mg administered PO QD beginning Cycle 1 Day 1 until disease progression or unacceptable toxicity. Lenalidomide 10 mg administered PO QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity. Rituximab 375 mg/m^2 administered IV on Day 1 of each 28-day cycle for 6 cycles.
  Interventions: Drug: Ibrutinib; Drug: Lenalidomide; Drug: Rituximab
- Phase 1b: Enrolled at Lenalidomide Dose 15 mg (Dose Level 1+) (Experimental): Re-escalation cohort: Ibrutinib 560 mg administered PO QD beginning Cycle 1 Day 1 until disease progression or unacceptable toxicity. Lenalidomide 15 mg administered PO QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity. Rituximab 375 mg/m^2 administered IV on Day 1 of each 28-day cycle for 6 cycles.
  Interventions: Drug: Ibrutinib; Drug: Lenalidomide; Drug: Rituximab
- Phase 1b: Enrolled at Lenalidomide Dose 20 mg (Dose Level 2) (Experimental): Ibrutinib 560 mg administered PO QD beginning Cycle 1 Day 1 until disease progression or unacceptable toxicity. Lenalidomide 20 mg administered PO QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity. Rituximab 375 mg/m^2 administered IV on Day 1 of each 28-day cycle for 6 cycles.
  Interventions: Drug: Ibrutinib; Drug: Lenalidomide; Drug: Rituximab
- Phase 1b: Enrolled at Lenalidomide Dose 25 mg (Dose Level 3) (Experimental): Ibrutinib 560 mg administered PO QD beginning Cycle 1 Day 1 until disease progression or unacceptable toxicity. Lenalidomide 25 mg administered PO QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity. Rituximab 375 mg/m^2 administered IV on Day 1 of each 28-day cycle for 6 cycles.
  Interventions: Drug: Ibrutinib; Drug: Lenalidomide; Drug: Rituximab
- Phase 2: Enrolled at Lenalidomide Dose 20 mg (Experimental): Ibrutinib 560 mg administered PO QD beginning Cycle 1 Day 1 until disease progression or unacceptable toxicity. Lenalidomide 20 mg administered PO QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity. Rituximab 375 mg/m^2 administered IV on Day 1 of each 28-day cycle for 6 cycles.
  Interventions: Drug: Ibrutinib; Drug: Lenalidomide; Drug: Rituximab
- Phase 2: Enrolled at Lenalidomide Dose 25 mg (Experimental): Ibrutinib 560 mg administered PO QD beginning Cycle 1 Day 1 until disease progression or unacceptable toxicity. Lenalidomide 25 mg administered PO QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity. Rituximab 375 mg/m^2 administered IV on Day 1 of each 28-day cycle for 6 cycles.
  Interventions: Drug: Ibrutinib; Drug: Lenalidomide; Drug: Rituximab

INTERVENTIONS:
Drug: Ibrutinib
Drug: Lenalidomide
Drug: Rituximab

SUMMARY:
This Phase 1b/2 study is designed to assess the safety and efficacy of ibrutinib in combination with lenalidomide and rituximab in subjects with relapsed/refractory diffuse large B-cell lymphoma (DLBCL) not eligible for transplant.

DETAILED DESCRIPTION:
Phase 1b: In the dose escalation portion of the study, various cohorts with escalating doses of lenalidomide may be explored, using the 3+3+3 principle for dose determination.

Phase 2: This will be conducted as an international, multicenter, open-label study. Eligible subjects will receive ibrutinib, lenalidomide and rituximab.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed relapsed/ refractory DLBCL
* Must have previously received first line treatment regimen
* Must be ineligible for high dose therapy/ stem cell transplantation
* Measurable disease sites on computed tomography (CT) scan (>1.5 cm in longest dimension)
* prothrombin time/international normalized ratio (PT/INR) < 1.5 x upper limit of normal (ULN) and partial thromboplastin time (PTT; activated partial thromboplastin time [aPTT]) <1.5 x ULN
* Men and women ≥18 years of age
* Eastern Cooperative Oncology Group (ECOG) < 2
* Adequate hepatic and renal function
* Adequate hematologic function

Exclusion Criteria:

* Medically apparent central nervous system lymphoma or leptomeningeal disease
* History of allogeneic stem-cell (or other organ) transplantation
* Any chemotherapy, external beam radiation therapy, or anticancer antibodies within 2 weeks
* Radio- or toxin-immunoconjugates within 10 weeks
* Concurrent enrollment in another therapeutic investigational study or have previously taken ibrutinib and/or lenalidomide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2014-03-13 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jutta K. Neuenburg, MD, PhD, Study Director — Pharmacyclics LLC.
Locations (40):
- United States (22):
  - University of Alabama, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Cedar Sinai Medical Center, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Tulane Medical Center, New Orleans, Louisiana
  - Karmanos Cancer Institute, Detroit, Michigan
  - Comprehensive Cancer Center of Nevada, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Summit Medical Group, Morristown, New Jersey
  - Weill Cornell Medical Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - University of Cincinnati Health Barrett Center, Cincinnati, Ohio
  - Mid-Ohio Oncology/ Hematology, Columbus, Ohio
  - University of TN Medical Center, Knoxville, Tennessee
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - Baylor Charles Sammons Cancer Center, Dallas, Texas
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Medical Oncology Associates, PS, Spokane, Washington
  - Northwest Medical Specialities, PLLC, Tacoma, Washington
- Belgium (5):
  - Ziekenhuis Netwerk Antwerpen - Campus Stuivenberg, Antwerp
  - CHU Brugmann, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
- Germany (4):
  - Universiaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Klinikum der Universitaet Muenchen - Campus Grosshadern, Munich, Bavaria
  - Klinikum rechts der Isar - Technische Universitaet Muenchen, III. Medizinische Klinik und Polyklinik, Munich, Bavaria
  - Universitaetsklinikum Wuerzburg, Medizinische Klinik und Poliklinik II, Würzburg, Bavaria
- United Kingdom (9):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - University Hospital of Wales, Cardiff
  - Northwick Park Hospital, Harrow
  - The Leeds Teaching Hospitals, Leeds
  - Kings College Hospital, London
  - University College London Hospitals, London
  - The Christie NHS Foundation Trust, Manchester
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - The Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Requests for access to individual participant data from clinical studies conducted by Pharmacyclics LLC, an AbbVie Company, can be submitted through Yale Open Data Access (YODA) Project site at the following link.
URL: http://yoda.yale.edu

REFERENCES:
- [Derived] Ramchandren R, Johnson P, Ghosh N, Ruan J, Ardeshna KM, Johnson R, Verhoef G, Cunningham D, de Vos S, Kassam S, Fayad L, Radford J, Bailly S, Offner F, Morgan D, Munoz J, Ping J, Szafer-Glusman E, Eckert K, Neuenburg JK, Goy A. The iR2 regimen (ibrutinib plus lenalidomide and rituximab) for relapsed/refractory DLBCL: A multicentre, non-randomised, open-label phase 2 study. EClinicalMedicine. 2022 Dec 26;56:101779. doi: 10.1016/j.eclinm.2022.101779. eCollection 2023 Feb. PMID 36618900
- [Derived] Goy A, Ramchandren R, Ghosh N, Munoz J, Morgan DS, Dang NH, Knapp M, Delioukina M, Kingsley E, Ping J, Beaupre DM, Neuenburg JK, Ruan J. Ibrutinib plus lenalidomide and rituximab has promising activity in relapsed/refractory non-germinal center B-cell-like DLBCL. Blood. 2019 Sep 26;134(13):1024-1036. doi: 10.1182/blood.2018891598. Epub 2019 Jul 22. PMID 31331917

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants had relapsed/refractory diffuse large B-cell lymphoma (DLBCL). In the Phase 1b portion of the study, all subtypes of DLBCL and participants with transformed disease were enrolled. In the Phase 2 portion of the study, only participants with non-germinal-center B-cell-like (non-GCB) DLBCL were enrolled.
Pre-assignment Details: In the Phase 1b portion of this study, different dose levels of lenalidomide were explored, and dose escalation of lenalidomide followed the 3+3+3 dose escalation schema.
  A total of 138 participants enrolled in the study; however, 4 participants exited the study without receiving any treatment, and are not presented in any data table.
Period: Overall Study
Arm/Group | Phase 1b: Enrolled at Lenalidomide Dose 15 mg (Dose Level 1) | Phase 1b: Enrolled at Lenalidomide Dose 10 mg (Dose Level -1) | Phase 1b: Enrolled at Lenalidomide Dose 15 mg (Dose Level 1+) | Phase 1b: Enrolled at Lenalidomide Dose 20 mg (Dose Level 2) | Phase 1b: Enrolled at Lenalidomide Dose 25 mg (Dose Level 3) | Phase 2: Enrolled at Lenalidomide Dose 20 mg | Phase 2: Enrolled at Lenalidomide Dose 25 mg
Started | 12 | 7 | 9 | 9 | 8 | 55 | 34
Completed (Participants remained on study until disease progression or unacceptable toxicity. "Reason Not Completed" rows display participants' primary reason for exiting the study.) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 12 | 7 | 9 | 9 | 8 | 55 | 34
Not completed — Death | 6 | 7 | 5 | 6 | 4 | 32 | 22
Not completed — Study Closure by Sponsor | 3 | 0 | 2 | 2 | 2 | 12 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 1 | 1 | 1 | 3 | 0
Not completed — Other, Not Specified | 0 | 0 | 1 | 0 | 1 | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Phase 1: Enrolled at Lenalidomide Dose 15 mg (Dose Level 1); Phase 1: Enrolled at Lenalidomide Dose 15 mg (Dose Level 1+): Ibrutinib 560 mg administered PO QD beginning Cycle 1 Day 1 until disease progression or unacceptable toxicity. Lenalidomide 15 mg administered PO QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity. Rituximab 375 mg/m^2 administered IV on Day 1 of each 28-day cycle for 6 cycles.
- Phase 1: Enrolled at Lenalidomide Dose 10 mg (Dose Level -1): Ibrutinib 560 mg administered PO QD beginning Cycle 1 Day 1 until disease progression or unacceptable toxicity. Lenalidomide 10 mg administered PO QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity. Rituximab 375 mg/m^2 administered intravenously (IV) on Day 1 of each 28-day cycle for 6 cycles.
- Phase 1: Enrolled at Lenalidomide Dose 20 mg (Dose Level 2); Phase 2: Enrolled at Lenalidomide Dose 20 mg: Ibrutinib 560 mg administered PO QD beginning Cycle 1 Day 1 until disease progression or unacceptable toxicity. Lenalidomide 20 mg administered PO QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity. Rituximab 375 mg/m^2 administered IV on Day 1 of each 28-day cycle for 6 cycles.
- Phase 1: Enrolled at Lenalidomide Dose 25 mg (Dose Level 3); Phase 2: Enrolled at Lenalidomide Dose 25 mg: Ibrutinib 560 mg administered PO QD beginning Cycle 1 Day 1 until disease progression or unacceptable toxicity. Lenalidomide 25 mg administered PO QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity. Rituximab 375 mg/m^2 administered IV on Day 1 of each 28-day cycle for 6 cycles.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Enrolled at Lenalidomide Dose 15 mg (Dose Level 1) | Phase 1: Enrolled at Lenalidomide Dose 10 mg (Dose Level -1) | Phase 1: Enrolled at Lenalidomide Dose 15 mg (Dose Level 1+) | Phase 1: Enrolled at Lenalidomide Dose 20 mg (Dose Level 2) | Phase 1: Enrolled at Lenalidomide Dose 25 mg (Dose Level 3) | Phase 2: Enrolled at Lenalidomide Dose 20 mg | Phase 2: Enrolled at Lenalidomide Dose 25 mg | Total
Number analyzed (Participants) | 12 | 7 | 9 | 9 | 8 | 55 | 34 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (13.13) | 58.4 (7.63) | 65.3 (13.44) | 66.0 (8.63) | 62.9 (14.23) | 63.1 (11.75) | 64.9 (12.52) | 63.9 (11.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 5 | 5 | 3 | 23 | 14 | 57
  Male | 8 | 4 | 4 | 4 | 5 | 32 | 20 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 1 | 0 | 0 | 0 | 5 | 10
  Not Hispanic or Latino | 11 | 4 | 8 | 9 | 8 | 55 | 29 | 124
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
  Black or African American | 1 | 1 | 1 | 0 | 1 | 2 | 1 | 7
  White | 11 | 5 | 8 | 9 | 7 | 51 | 30 | 121
  Multiple Races | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Declined to Answer/Unknown | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Recommended Phase 2 Dose of Lenalidomide in Combination With Fixed Doses of Ibrutinib and Rituximab in Participants With Relapsed or Refractory Diffuse Large B Cell Lymphoma (DLBCL)
Description: The dose levels of lenalidomide were explored, and dose escalation of lenalidomide followed the 3+3+3 dose escalation schema. A Dose Level Review Committee evaluated safety data following completion of each dose observation period of the Phase 1b portion.
Time Frame: Estimated median time on study in Phase 1b was 59.6 months.
Population: All-Treated Analysis Population (Phase 1b): participants who received any dose of study drug(s).
Measure: Number; unit: mg
Groups:
- All Phase 1b Participants: Ibrutinib 560 mg administered PO QD beginning Cycle 1 Day 1 until disease progression or unacceptable toxicity. Lenalidomide 10, 15, 20, or 25 mg administered PO QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity. Rituximab 375 mg/m^2 administered IV on Day 1 of each 28-day cycle for 6 cycles.
Arm/Group | All Phase 1b Participants
Number analyzed (Participants) | 45
mg | 20

2. Primary Outcome: Phase 1b: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, and Discontinuations Due to TEAEs
Description: An adverse event (AE) is any untoward medical occurrence, which does not necessarily have a causal relationship with treatment. A serious AE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires in-patient hospitalization > 24 hours or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is an important medical event. AEs that started or worsened during the treatment-emergent period and all possibly related or related AEs were considered TEAEs. Related events were those that were considered possibly related or related to study drug per investigator's judgment. Events were graded per the national Cancer Institute's Common Terminology Criteria for Adverse Events, version 4.03: Grade 1=mild; grade 2=moderate; grade 3=severe; grade 4=life-threatening; grade 5=death.
Time Frame: From first dose of study drug up to 30 days after last dose of study drug. Phase 1b median duration of ibrutinib exposure was 4.4 months; median duration of lenalidomide exposure was 4.4 months; median total number of doses of rituximab received was 4.0.
Population: All-Treated Analysis Population (Phase 1): participants who received any dose of study drug(s).
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b: Enrolled at Lenalidomide Dose 15 mg (Dose Level 1); Phase 1b: Enrolled at Lenalidomide Dose 15 mg (Dose Level 1+): Ibrutinib 560 mg administered PO QD beginning Cycle 1 Day 1 until disease progression or unacceptable toxicity. Lenalidomide 15 mg administered PO QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity. Rituximab 375 mg/m^2 administered IV on Day 1 of each 28-day cycle for 6 cycles.
- Phase 1b: Enrolled at Lenalidomide Dose 10 mg (Dose Level -1): Ibrutinib 560 mg administered PO QD beginning Cycle 1 Day 1 until disease progression or unacceptable toxicity. Lenalidomide 10 mg administered PO QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity. Rituximab 375 mg/m^2 administered intravenously (IV) on Day 1 of each 28-day cycle for 6 cycles.
Arm/Group | Phase 1b: Enrolled at Lenalidomide Dose 15 mg (Dose Level 1) | Phase 1b: Enrolled at Lenalidomide Dose 10 mg (Dose Level -1) | Phase 1b: Enrolled at Lenalidomide Dose 15 mg (Dose Level 1+) | Phase 1b: Enrolled at Lenalidomide Dose 20 mg (Dose Level 2) | Phase 1b: Enrolled at Lenalidomide Dose 25 mg (Dose Level 3)
Number analyzed (Participants) | 12 | 7 | 9 | 9 | 8
Participants
  Any TEAE | 12 | 7 | 9 | 9 | 8
  Any Grade >=3 TEAE | 11 | 6 | 9 | 9 | 7
  Any Study Drug-Related TEAE | 12 | 5 | 9 | 8 | 8
  Any Grade >=3 Study Drug-Related TEAE | 10 | 3 | 8 | 7 | 7
  Any Ibrutinib-Related TEAE | 12 | 5 | 9 | 8 | 8
  Any Grade >=3 Ibrutinib-Related TEAE | 10 | 3 | 7 | 7 | 6
  Any Lenalidomide-Related TEAE | 12 | 5 | 9 | 8 | 8
  Any Grade >=3 Lenalidomide-Related TEAE | 9 | 3 | 8 | 7 | 6
  Any Rituximab-Related TEAE | 6 | 4 | 7 | 6 | 7
  Any Grade >= 3 Rituximab-Related TEAE | 1 | 2 | 7 | 5 | 3
  Any TEAE Leading to Dose Reduction of Any Study Drug | 4 | 0 | 4 | 4 | 5
  Any TEAE Leading to Dose Reduction of Ibrutinib | 3 | 0 | 4 | 3 | 3
  Any TEAE Leading to Dose Reduction of Lenalidomide | 2 | 0 | 3 | 4 | 4
  Any TEAE Leading to Dose Delay of Any Study Drug | 6 | 4 | 7 | 8 | 8
  Any TEAE Leading to Dose Delay of Ibrutinib | 6 | 4 | 7 | 8 | 8
  Any TEAE Leading to Dose Delay of Lenalidomide | 6 | 3 | 7 | 7 | 8
  Any TEAE Leading to Dose Delay of Rituximab | 4 | 1 | 6 | 4 | 4
  Any TEAE Leading to Discontinuation of Any Study Drug | 4 | 2 | 3 | 2 | 1
  Any TEAE Leading to Discontinuation of Ibrutinib Dose | 4 | 2 | 3 | 2 | 1
  Any TEAE Leading to Discontinuation of Lenalidomide Dose | 4 | 2 | 3 | 2 | 1
  Any TEAE Leading to Discontinuation of Rituximab Dose | 3 | 2 | 3 | 2 | 1
  Any Serious TEAE | 4 | 6 | 7 | 5 | 6
  Any Grade >=3 Serious TEAE | 4 | 6 | 6 | 4 | 6
  Any Treatment-Related Serious TEAE | 0 | 2 | 4 | 2 | 3
  Any Ibrutinib-Related Serious TEAE | 0 | 2 | 4 | 2 | 3
  Any Lenalidomide-Related Serious TEAE | 0 | 2 | 4 | 2 | 3
  Any Rituximab-Related Serious TEAE | 0 | 2 | 2 | 1 | 0
  Any Fatal TEAE | 0 | 2 | 2 | 1 | 1

3. Primary Outcome: Phase 2: Overall Response Rate (ORR)
Description: The ORR was defined as the percentage of participants who achieve either a partial response (PR) or complete response (CR), according to the Revised International Working Group Response Criteria for Malignant Lymphoma or Lugano Classification (Cheson 2014), as assessed by the investigator in response-evaluable population. The 95% confidence interval (CI) was calculated using the exact method.
Time Frame: Estimated median time on study in Phase 2 was 35.0 months.
Population: Response-Evaluable Population: participants who had measurable disease at baseline and had at least 1 adequate post-treatment disease assessment by the investigator.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 2 Total: Enrolled at Lenalidomide Dose 20 or 25 mg: Ibrutinib 560 mg administered PO QD beginning Cycle 1 Day 1 until disease progression or unacceptable toxicity. Lenalidomide 20 or 25 mg administered PO QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity. Rituximab 375 mg/m^2 administered IV on Day 1 of each 28-day cycle for 6 cycles.
Arm/Group | Phase 2: Enrolled at Lenalidomide Dose 20 mg | Phase 2: Enrolled at Lenalidomide Dose 25 mg | Phase 2 Total: Enrolled at Lenalidomide Dose 20 or 25 mg
Number analyzed (Participants) | 53 | 32 | 85
percentage of participants | 52.8 [38.6 to 66.7] | 43.8 [26.4 to 62.3] | 49.4 [38.4 to 60.5]

4. Secondary Outcome: Phase 1b: ORR
Description: The ORR was defined as the percentage of participants who achieve either a PR or CR, according to the Revised International Working Group Response Criteria for Malignant Lymphoma (Cheson 2007), as assessed by the Investigator in response-evaluable population, where CR=disappearance of all evidence of disease and PR=regression of measurable disease and no new sites. The 95% CI was calculated using the exact method.
Time Frame: Estimated median time on study in Phase 1b was 59.6 months.
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 1b: Enrolled at Lenalidomide Dose 10 mg (Dose Level -1): Ibrutinib 560 mg administered PO QD beginning Cycle 1 Day 1 until disease progression or unacceptable toxicity. Lenalidomide 10 mg administered PO QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity. Rituximab 375 mg/m^2 administered IV on Day 1 of each 28-day cycle for 6 cycles.
- Phase 1b Total: Enrolled at Lenalidomide Dose 10 to 25 mg (All Dose Levels): Ibrutinib 560 mg administered PO QD beginning Cycle 1 Day 1 until disease progression or unacceptable toxicity. Lenalidomide 10, 15, 20, or 25 mg administered PO QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity. Rituximab 375 mg/m^2 administered IV on Day 1 of each 28-day cycle for 6 cycles.
Arm/Group | Phase 1b: Enrolled at Lenalidomide Dose 15 mg (Dose Level 1) | Phase 1b: Enrolled at Lenalidomide Dose 10 mg (Dose Level -1) | Phase 1b: Enrolled at Lenalidomide Dose 15 mg (Dose Level 1+) | Phase 1b: Enrolled at Lenalidomide Dose 20 mg (Dose Level 2) | Phase 1b: Enrolled at Lenalidomide Dose 25 mg (Dose Level 3) | Phase 1b Total: Enrolled at Lenalidomide Dose 10 to 25 mg (All Dose Levels)
Number analyzed (Participants) | 9 | 7 | 7 | 9 | 8 | 40
percentage of participants | 44.4 [13.7 to 78.8] | 0 [0 to 41.0] | 71.4 [29.0 to 96.3] | 22.2 [2.8 to 60.0] | 75.0 [34.9 to 96.8] | 42.5 [27.0 to 59.1]

5. Secondary Outcome: Phase 1b: Complete Response (CR) Rate
Description: The CR rate was defined as the percentage of participants who achieve a CR, according to the Revised International Working Group Response Criteria for Malignant Lymphoma (Cheson 2007), as assessed by the Investigator in response-evaluable population, where CR=disappearance of all evidence of disease, as assessed by the Investigator.
Time Frame: Estimated median time on Phase 1b study was 59.6 months.
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1b: Enrolled at Lenalidomide Dose 15 mg (Dose Level 1) | Phase 1b: Enrolled at Lenalidomide Dose 10 mg (Dose Level -1) | Phase 1b: Enrolled at Lenalidomide Dose 15 mg (Dose Level 1+) | Phase 1b: Enrolled at Lenalidomide Dose 20 mg (Dose Level 2) | Phase 1b: Enrolled at Lenalidomide Dose 25 mg (Dose Level 3) | Phase 1b Total: Enrolled at Lenalidomide Dose 10 to 25 mg (All Dose Levels)
Number analyzed (Participants) | 9 | 7 | 7 | 9 | 8 | 40
percentage of participants | 33.3 | 0 | 42.9 | 11.1 | 50.0 | 27.5

6. Secondary Outcome: Phase 2: CR Rate
Description: The CR rate was defined as the percentage of participants who achieve a CR, according to the Revised International Working Group Response Criteria for Malignant Lymphoma or Lugano Classification (see Cheson, 2014 for detailed criteria) in response-evaluable population, as assessed by the Investigator.
Time Frame: Estimated median time on study in Phase 2 was 35.0 months.
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Enrolled at Lenalidomide Dose 20 mg | Phase 2: Enrolled at Lenalidomide Dose 25 mg | Phase 2 Total: Enrolled at Lenalidomide Dose 20 or 25 mg
Number analyzed (Participants) | 53 | 32 | 89
percentage of participants | 32.1 | 21.9 | 28.2

7. Secondary Outcome: Phase 2: Duration of Response (DOR)
Description: DOR is defined as the time from the date of the first documented response (CR or PR) to the first documented evidence of disease progression (PD) according to the Revised International Working Group Response Criteria for Malignant Lymphoma or Lugano Classification (Cheson 2014) or death from any cause. For participants who had achieved an overall response but did not die or progress at the time of analysis, DOR was censored on the date of the last adequate post-baseline disease assessment, or on the date of the first occurrence of response (CR or PR) if there was no disease assessment afterwards. 2-sided 95% CI is estimated by Kaplan-Meier method.
Time Frame: Estimated median time on study in Phase 2 was 35.0 months.
Population: All-Treated Analysis Population (Phase 2): participants who received any dose of study drug(s). Participant who achieved Overall Response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Enrolled at Lenalidomide Dose 20 mg | Phase 2: Enrolled at Lenalidomide Dose 25 mg | Phase 2 Total: Enrolled at Lenalidomide Dose 20 or 25 mg
Number analyzed (Participants) | 28 | 14 | 42
months | 38.3 [3.7 to NA] — The upper confidence limit is not estimable per the Brookmeyer and Crowley (1982) method. | 28.6 [2.8 to 28.6] | 38.3 [9.5 to NA] — The upper confidence limit is not estimable per the Brookmeyer and Crowley (1982) method.

8. Secondary Outcome: Phase 2: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of the first dose of study drug to confirmed PD according to the Revised International Working Group Response Criteria for Malignant Lymphoma or Lugano Classification (Cheson 2014) or death from any cause, whichever occurred first. For participants without disease progression or death, PFS data was censored at the date of the last tumor assessment. 2 sided 95% CI is estimated by Kaplan-Meier method.
Time Frame: Estimated median time on study in Phase 2 was 35.0 months.
Population: All-Treated Analysis Population (Phase 2): participants who received any dose of study drug(s).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Enrolled at Lenalidomide Dose 20 mg | Phase 2: Enrolled at Lenalidomide Dose 25 mg | Phase 2 Total: Enrolled at Lenalidomide Dose 20 or 25 mg
Number analyzed (Participants) | 55 | 34 | 89
months | 5.4 [3.4 to 11.3] | 4.7 [2.6 to 24.8] | 5.4 [3.4 to 6.3]

9. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS is defined as the time from the date of the first dose of study drug to the date of death due to any cause. For participants not known to have died at or prior to the database lock date, OS data was censored at the date last known alive. Participants who withdrew consent prior to study closure were censored on the date of the consent withdrawal. 2-sided 95% CI was estimated by Kaplan-Meier method.
Time Frame: Estimated median time on study in Phase 2 was 35.0 months.
Population: All-Treated Analysis Population (Phase 2): participants who received any dose of study drug(s).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Enrolled at Lenalidomide Dose 20 mg | Phase 2: Enrolled at Lenalidomide Dose 25 mg | Phase 2 Total: Enrolled at Lenalidomide Dose 20 or 25 mg
Number analyzed (Participants) | 55 | 34 | 89
months | 14.7 [9.7 to 32.8] | 11.6 [5.7 to NA] — The upper confidence limit is not estimable per the Brookmeyer and Crowley (1982) method. | 14.2 [9.7 to 28.1]

10. Secondary Outcome: Phase 2: Number of Participants With TEAEs, Serious TEAEs, and Discontinuations Due to TEAEs
Description: as for outcome 2
Time Frame: From first dose of study drug up to 30 days after last dose of study drug. Phase 2 median duration of ibrutinib exposure was 4.9 months; median duration of lenalidomide exposure was 4.7 months; median total number of doses of rituximab received was 5.0.
Population: All-Treated Analysis Population (Phase 2): participants who received any dose of study drug(s).
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2 Total: Enrolled at Lenalidomide Dose 20 or 25 mg: Ibrutinib 560 mg administered PO QD beginning Cycle 1 Day 1 until disease progression or unacceptable toxicity. Lenalidomide 20 to 25 mg administered PO QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity. Rituximab 375 mg/m^2 administered IV on Day 1 of each 28-day cycle for 6 cycles.
Arm/Group | Phase 2: Enrolled at Lenalidomide Dose 20 mg | Phase 2: Enrolled at Lenalidomide Dose 25 mg | Phase 2 Total: Enrolled at Lenalidomide Dose 20 or 25 mg
Number analyzed (Participants) | 55 | 34 | 89
Participants
  Any TEAE | 55 | 34 | 89
  Any Grade >=3 TEAE | 51 | 30 | 81
  Any Study Drug-Related TEAE | 52 | 33 | 85
  Any Grade >=3 Study Drug-Related TEAE | 41 | 25 | 66
  Any Ibrutinib-Related TEAE | 50 | 32 | 82
  Any Grade >=3 Ibrutinib-Related TEAE | 36 | 24 | 60
  Any Lenalidomide-Related TEAE | 51 | 32 | 83
  Any Grade >=3 Lenalidomide-Related TEAE | 40 | 25 | 65
  Any Rituximab-Related TEAE | 37 | 25 | 62
  Any Grade >= 3 Rituximab-Related TEAE | 18 | 13 | 31
  Any TEAE Leading to Dose Reduction of Any Study Drug | 23 | 14 | 37
  Any TEAE Leading to Dose Reduction of Ibrutinib | 12 | 9 | 21
  Any TEAE Leading to Dose Reduction of Lenalidomide | 21 | 14 | 35
  Any TEAE Leading to Dose Delay of Any Study Drug | 40 | 29 | 69
  Any TEAE Leading to Dose Delay of Ibrutinib | 38 | 28 | 66
  Any TEAE Leading to Dose Delay of Lenalidomide | 37 | 26 | 63
  Any TEAE Leading to Dose Delay of Rituximab | 10 | 6 | 16
  Any TEAE Leading to Discontinuation of Any Study Drug | 11 | 7 | 18
  Any TEAE Leading to Discontinuation of Ibrutinib Dose | 11 | 5 | 16
  Any TEAE Leading to Discontinuation of Lenalidomide Dose | 11 | 7 | 18
  Any TEAE Leading to Discontinuation of Rituximab Dose | 6 | 4 | 10
  Any Serious TEAE | 32 | 25 | 57
  Any Grade >=3 Serious TEAE | 29 | 21 | 50
  Any Treatment-Related Serious TEAE | 16 | 12 | 28
  Any Ibrutinib-Related Serious TEAE | 14 | 12 | 26
  Any Lenalidomide-Related Serious TEAE | 16 | 10 | 26
  Any Rituximab-Related Serious TEAE | 4 | 5 | 9
  Any Fatal TEAE | 8 | 4 | 12

ADVERSE EVENTS:
Time Frame: All Cause Mortality Time Frame: Estimated median time on study in Phase 1b was 59.6 months. Estimated median time on study in Phase 2 was 35.0 months.
Description: Adverse Events Time Frame: From first dose of study drug up to 30 days after last dose of study drug. Phase 1b median duration of ibrutinib exposure was 4.4 months; median duration of lenalidomide exposure was 4.4 months; median total number of doses of rituximab received was 4.0. Phase 2 median duration of ibrutinib exposure was 4.9 months; median duration of lenalidomide exposure was 4.7 months; median total number of doses of rituximab received was 5.0.
Arm/Group | Phase 1b: Enrolled at Lenalidomide Dose 15 mg (Dose Level 1) | Phase 1b: Enrolled at Lenalidomide Dose 10 mg (Dose Level -1) | Phase 1b: Enrolled at Lenalidomide Dose 15 mg (Dose Level 1+) | Phase 1b: Enrolled at Lenalidomide Dose 20 mg (Dose Level 2) | Phase 1b: Enrolled at Lenalidomide Dose 25 mg (Dose Level 3) | Phase 2: Enrolled at Lenalidomide Dose 20 mg | Phase 2: Enrolled at Lenalidomide Dose 25 mg
All-Cause Mortality (participants affected / at risk) | 7/12 | 7/7 | 5/9 | 7/9 | 5/8 | 33/55 | 22/34
Serious Adverse Events (participants affected / at risk) | 4/12 | 6/7 | 7/9 | 5/9 | 6/8 | 32/55 | 25/34
Other Adverse Events (participants affected / at risk) | 12/12 | 7/7 | 9/9 | 9/9 | 8/8 | 54/55 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b: Enrolled at Lenalidomide Dose 15 mg (Dose Level 1) (N=12) | Phase 1b: Enrolled at Lenalidomide Dose 10 mg (Dose Level -1) (N=7) | Phase 1b: Enrolled at Lenalidomide Dose 15 mg (Dose Level 1+) (N=9) | Phase 1b: Enrolled at Lenalidomide Dose 20 mg (Dose Level 2) (N=9) | Phase 1b: Enrolled at Lenalidomide Dose 25 mg (Dose Level 3) (N=8) | Phase 2: Enrolled at Lenalidomide Dose 20 mg (N=55) | Phase 2: Enrolled at Lenalidomide Dose 25 mg (N=34)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 2 (2)
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (4) | 1 (1) | 1 (2)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
GASTROSPLENIC FISTULA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
INCARCERATED INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CATHETER SITE PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHILLS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 5 (5) | 4 (4)
BILE DUCT STENOSIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GALLBLADDER ENLARGEMENT (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACUTE SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CANDIDA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 2 (3) | 2 (2) | 1 (1)
CELLULITIS ORBITAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ESCHERICHIA SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FOLLICULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATOMA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LYMPHANGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NEUTROPENIC SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PERITONITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SALMONELLA BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (4) | 0 (0)
WOUND SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
MOBILITY DECREASED (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
BOWEN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 5 (5) | 3 (3)
INTRADUCTAL PROLIFERATIVE BREAST LESION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OCULAR LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EMBOLIC CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DELIRIUM (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PROSTATIC OBSTRUCTION (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PURPURA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b: Enrolled at Lenalidomide Dose 15 mg (Dose Level 1) (N=12) | Phase 1b: Enrolled at Lenalidomide Dose 10 mg (Dose Level -1) (N=7) | Phase 1b: Enrolled at Lenalidomide Dose 15 mg (Dose Level 1+) (N=9) | Phase 1b: Enrolled at Lenalidomide Dose 20 mg (Dose Level 2) (N=9) | Phase 1b: Enrolled at Lenalidomide Dose 25 mg (Dose Level 3) (N=8) | Phase 2: Enrolled at Lenalidomide Dose 20 mg (N=55) | Phase 2: Enrolled at Lenalidomide Dose 25 mg (N=34)
ANAEMIA (Blood and lymphatic system disorders) | 4 (6) | 0 (0) | 3 (6) | 3 (22) | 2 (6) | 17 (88) | 11 (16)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INCREASED TENDENCY TO BRUISE (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 2 (3) | 0 (0) | 2 (2) | 8 (13) | 5 (6)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (7) | 0 (0) | 0 (0) | 1 (4) | 1 (2) | 3 (35) | 3 (6)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPHOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 5 (13) | 0 (0) | 6 (46) | 3 (22) | 5 (41) | 25 (126) | 14 (68)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SPONTANEOUS HAEMATOMA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 (8) | 2 (5) | 4 (9) | 4 (21) | 3 (10) | 11 (61) | 10 (36)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
PALPITATIONS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 4 (4)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
DEAFNESS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
HYPOACUSIS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
CHALAZION (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRY AGE-RELATED MACULAR DEGENERATION (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DRY EYE (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (7) | 6 (8)
EXOPHTHALMOS (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EYE OEDEMA (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYE PAIN (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
EYE PRURITUS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
LACRIMATION INCREASED (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
METAMORPHOPSIA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OCULAR HYPERAEMIA (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OPTIC NERVE COMPRESSION (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIORBITAL SWELLING (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHOTOPHOBIA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TRICHIASIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
VISUAL ACUITY REDUCED (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VISUAL IMPAIRMENT (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 9 (11) | 7 (10)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (2)
CONSTIPATION (Gastrointestinal disorders) | 5 (5) | 2 (2) | 4 (4) | 4 (4) | 3 (5) | 11 (17) | 10 (13)
DEFAECATION URGENCY (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 9 (22) | 3 (4) | 3 (3) | 4 (8) | 7 (16) | 32 (83) | 13 (29)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 8 (9) | 8 (8)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 7 (7) | 3 (3)
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FAECES DISCOLOURED (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 5 (9) | 1 (1)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GINGIVAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
GINGIVAL SWELLING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GLOSSODYNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
HYPERCHLORHYDRIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MELAENA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
MOUTH ULCERATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 7 (10) | 3 (4) | 3 (4) | 3 (5) | 4 (8) | 17 (20) | 9 (15)
ORAL DISORDER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 2 (2)
PARAESTHESIA ORAL (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SALIVARY GLAND CALCULUS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 7 (7) | 5 (17)
TONGUE ULCERATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TOOTH LOSS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 3 (6) | 2 (3) | 12 (19) | 5 (8)
ADVERSE DRUG REACTION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (2) | 4 (4)
CHEST DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
CHILLS (General disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
FACE OEDEMA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 6 (8) | 3 (3) | 5 (9) | 2 (3) | 3 (4) | 22 (34) | 16 (22)
GAIT DISTURBANCE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
INFUSION SITE EXTRAVASATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFUSION SITE SWELLING (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MALAISE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 3 (3) | 3 (3)
NODULE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 2 (2) | 1 (1) | 3 (3) | 3 (3) | 4 (5) | 21 (30) | 8 (10)
PAIN (General disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 2 (2)
PERIPHERAL SWELLING (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 4 (4)
PYREXIA (General disorders) | 0 (0) | 1 (2) | 2 (4) | 0 (0) | 3 (3) | 2 (2) | 3 (3)
VESSEL PUNCTURE SITE BRUISE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEPATIC CYST (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
HEPATOMEGALY (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
HYPOGAMMAGLOBULINAEMIA (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
SEASONAL ALLERGY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
ARTHRITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLISTER INFECTED (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
CHRONIC SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CLOSTRIDIUM COLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONJUNCTIVITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 4 (4) | 1 (1)
CONJUNCTIVITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
CORONAVIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CYSTITIS KLEBSIELLA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EYE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
FOLLICULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (3)
FUNGAL SKIN INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
FURUNCLE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IMPETIGO (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
NAIL INFECTION (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (10) | 1 (1)
ONYCHOMYCOSIS (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
OTITIS EXTERNA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 2 (2)
PSEUDOMONAS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PUSTULE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RASH PUSTULAR (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (7) | 2 (5)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINOVIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
SINUSITIS (Infections and infestations) | 1 (2) | 1 (2) | 2 (2) | 0 (0) | 1 (2) | 4 (5) | 4 (6)
SINUSITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TINEA PEDIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 2 (9) | 12 (22) | 4 (6)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 7 (8) | 2 (4)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WOUND ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WOUND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 6 (7) | 5 (8)
EYE CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
IMPACTED FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
LIMB INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MOUTH INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NAIL INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
SCRATCH (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN ABRASION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
WOUND (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (2) | 2 (3) | 1 (5)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (3)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
BLOOD CREATINE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (8) | 0 (0)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BLOOD URINE PRESENT (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BODY TEMPERATURE FLUCTUATION (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CARDIAC MURMUR (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
CREATININE RENAL CLEARANCE DECREASED (Investigations) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 3 (3) | 6 (11) | 6 (12)
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (2) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (7) | 7 (53) | 2 (2)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (14) | 2 (5)
STAPHYLOCOCCUS TEST POSITIVE (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
VITAMIN D DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 8 (11) | 4 (8)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 4 (7) | 2 (5) | 2 (3) | 8 (11) | 5 (7)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
ENZYME ABNORMALITY (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (6) | 0 (0) | 1 (5) | 2 (2) | 1 (5)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 3 (3) | 1 (1)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 1 (1)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 2 (2)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4 (8) | 1 (1) | 3 (7) | 3 (3) | 3 (6) | 16 (22) | 4 (7)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (4) | 2 (2) | 1 (6) | 11 (19) | 2 (2)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 2 (5) | 1 (1) | 1 (2)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
MALNUTRITION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 2 (4) | 2 (4) | 2 (2) | 9 (12) | 5 (7)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 2 (4) | 10 (12) | 4 (4)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 2 (2)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
MUSCLE ATROPHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2) | 2 (3) | 0 (0) | 3 (3) | 12 (18) | 7 (10)
MUSCLE TIGHTNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 6 (6)
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (4) | 4 (8) | 6 (8)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (5) | 1 (1) | 1 (1) | 5 (5) | 5 (8)
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APHASIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
ATAXIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BALANCE DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 4 (5) | 0 (0) | 2 (2) | 3 (5) | 1 (2) | 11 (16) | 7 (7)
DIZZINESS POSTURAL (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
DYSARTHRIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
HEAD DISCOMFORT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 3 (4) | 4 (6)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 2 (2)
PARKINSON'S DISEASE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0)
PERIPHERAL SENSORIMOTOR NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 11 (20) | 7 (14)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
RESTLESS LEGS SYNDROME (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
SPEECH DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (2)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
DISORIENTATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 2 (2)
IRRITABILITY (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
STRESS (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BLADDER TRABECULATION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 3 (11) | 1 (1)
URETHRAL STENOSIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
GENITAL RASH (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OEDEMA GENITAL (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
ALLERGIC SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 2 (4) | 0 (0) | 3 (5) | 18 (27) | 13 (19)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 3 (3)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (3) | 1 (2) | 3 (3) | 3 (3) | 17 (23) | 7 (9)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (7) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 5 (7) | 3 (4)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 4 (5) | 5 (5)
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NASAL SEPTUM PERFORATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 6 (9) | 1 (2)
PARANASAL SINUS HYPERSECRETION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 4 (7) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 4 (6) | 5 (5)
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (4) | 4 (4) | 3 (4)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
YAWNING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BLISTER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD BLISTER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 13 (15) | 7 (7)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (3)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 6 (9) | 2 (2)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MACULE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 4 (9) | 3 (3)
ONYCHOCLASIS (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PETECHIAE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 2 (3) | 5 (10) | 2 (3)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 7 (11) | 6 (8)
PURPURA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 7 (7)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 7 (11) | 3 (3)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 2 (5) | 1 (2) | 5 (11) | 3 (5) | 2 (3) | 15 (40) | 12 (35)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
SCAB (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN LESION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (4)
STASIS DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHYSICAL ASSAULT (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HOT FLUSH (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (3) | 1 (21) | 5 (15)
HYPOTENSION (Vascular disorders) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
PERIPHERAL COLDNESS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VARICOSE VEIN (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
1. Institution/Investigator will not publish without Sponsor prior review and approval
2. Institution/Investigator will not publish until the earlier of (i) results of study are submitted for publication (ii) notification that submission of the multicenter results are no longer planned (iii) 18 months after study termination.

DOCUMENTS (2):
  • Study Protocol (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT02077166/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT02077166/SAP_001.pdf